CLINICAL TRIAL: NCT01311986
Title: Chemokine Expression in Nummular Dermatitis and Atopic Dermatitis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Hsien-Ching Chiu, Department of Dermatology, National Taiwan University Hospital
Other Study IDs: 201006030R
Record Dates: First submitted 2011-03-08; First posted 2011-03-10 (Estimated); Last update posted 2011-04-22 (Estimated); Status verified 2011-03

CONDITIONS: Atopic Dermatitis; Nummular Eczema
Keywords: atopic dermatitis; nummular eczema; chemokines
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Patient serum, and epidermal keratinocytes for mRNA retrieval
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Patients with atopic dermatitis
- Patients with nummular eczema
- Normal control

SUMMARY:
The aim of this study is to measure the serum levels of CCL17, CCL18, CCL22 and CXCL10 and their expression levels in epidermis in AD and ND patients.

DETAILED DESCRIPTION:
Atopic dermatitis(AD) is a common cutaneous inflammatory disease. The pathogenesis of atopic dermatitis involves a complex interaction between atopy and environmental protein allergens which produces Th2 immune responses with IgE formation, Th2 cells dominate in lesions of atopic dermatitis, whereas Th1 and Th2 cells co-dominate in late eczematus lesions.

Nummular dermatitis(ND) is another common cutaneous inflammatory disease. The nummular patches and papules disseminated over four extremities and less over trunk . The serum levels of Th2 chemokines(CCL17, CCL22, CCL27) are elevated in AD patients. The expression levels of these chemokines in lesional epidermis are also increased. CCL18 which is derived from APC is also increased in the serum as well as lesional skin of AD patients. In contrast, there are very few reports regarding the chemokine expression profiles in ND patients. Because erosis is a remarkable exacerbating factor for ND. The investigators hypothesize that ND is a specialized contact dermatitis induced by environmental substances. It has been known, CCL17 and CXCL10 were highly expressed in lesion of allergic contant dermatitis, whereas almost no expression of these chemokines could be detected in lesions of irritant contact dermatitis.

The aim of this study is to measure the serum levels of CCL17, CCL18, CCL22 and CXCL10 and their expression levels in epidermis in AD and ND patients. The investigators hope that the results of this study will provide useful information for clinical differential diagnosis for AD and ND as well as understanding the pathogenesis of ND.

ELIGIBILITY:
Inclusion Criteria:

* age:20~40, atopic dermatitis, BSA>10%, no asthma
* age:20~40, nummular patches>10, no atopy

Exclusion Criteria:

* systemic immunosuppresive agents within 4 weeks
* high dose topical immunosuppresive agents within 4 weeks

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: patients with atopic dermatitis
  patients with nummular eczema without atopy
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-10 (Estimated); Study Completion 2012-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Hsien-Ching Chiu, MD, Principal Investigator — Department of Dermatology, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei, Taiwan